CLINICAL TRIAL: NCT02183220
Title: A Randomised, Double Blind, Placebo- and Active-controlled Parallel Group Study Investigating the Efficacy and Tolerability of Metamizol 0.5 g and 1.0 g in Patients With Episodic Moderate Tension Headache.
Brief Title: Efficacy and Tolerability of Metamizol in Patients With Episodic Moderate Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1093.16
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Dipyrone; Aspirin

ARMS (4):
- Metamizol high & Placebo (Experimental)
  Interventions: Drug: Metamizol; Drug: Metamizol placebo
- Metamizol low & Placebo (Experimental)
  Interventions: Drug: Metamizol; Drug: Metamizol placebo
- Acetylsalicylic acid & Placebo (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid (ASA); Drug: ASA placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Metamizol placebo; Drug: ASA placebo

INTERVENTIONS:
Drug: Metamizol
  Arms: Metamizol high & Placebo; Metamizol low & Placebo
Drug: Acetylsalicylic acid (ASA)
  Arms: Acetylsalicylic acid & Placebo
Drug: Metamizol placebo
  Arms: Metamizol high & Placebo; Metamizol low & Placebo; Placebo
Drug: ASA placebo
  Arms: Acetylsalicylic acid & Placebo; Placebo

SUMMARY:
The objective of the study was to evaluate the efficacy, safety and tolerability of a single peroral dose of 0.5 g and 1.0 g metamizol relative to placebo and 1.0 g acetylsalicylic acid in 2 episodes of moderate tension headache.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 65 years old
* Moderate episodic tension headache according to International Headache Society (I.H.S.) classification 2.1 (2.1.1 and 2.1.2) for at least one year
* At least two episodes of tension headache per month in the last three months prior to enrolment into this trial
* The episodes of tension headaches were usually treated by the patient successfully with a non-opioid-analgesic
* First episodic headache occurred at an age under 50 years
* Written informed consent according to Good Clinical Practice (GCP) and local regulations
* The patient was able to fill in the Patient's Diary

Exclusion Criteria:

* The patient usually needs for successful treatment of tension headache "Over The Counter" (OTC) analgesic in doses exceeding the doses tested here
* The patient takes an OTC-analgesic normally at the first signs of an episode of tension headache
* The patient has more than 15 episodes of tension headache per month
* Female patients whose episodic tension headache is strongly correlated with the start of hormonal contraception
* Concomitant treatment with (non-) prescriptional analgesics
* Pre- (less than 4 weeks prior to inclusion in this trial) and/or concomitant treatment with an antidepressive and/or antipsychotic drug
* Pre- (less than 2 weeks prior to inclusion in this trial) and/or concomitant treatment with any drug such as NSAIDs (Non-Steroidal Anti Inflammatory Drugs), propanolol, metroprolol, flunarizin, cyclandelate, valproic-acid, serotonergic antagonists, ergotamine, dihydroergotamines and benzodiazepines that may influence the headache symptomatology
* Use of benzodiazepines in the previous 24 hours to the administration of the study drug. Occasional use of benzodiazepines - up to 3 per week - is allowed
* Use of any drug with analgesic properties in the previous 24 hours to the administration of the study drug
* Concomitant treatment with any drug containing ASA and/or metamizol
* Concomitant treatment with anticoagulants such as heparin or coumarin-derivatives
* Alcohol and drug abuse according to DSM-IV (Diagnostic and Statistical Manual of Mental Disorders )
* Female patients in child-bearing age not using adequate means of birth control
* Pregnancy and/or lactation
* Gastrointestinal ulcers
* Liver and/or renal disease
* Bronchial asthma
* Relevant allergy or known hypersensitivity to the investigational drugs, its excipients and/or to other NSAIDs
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial
* Patients with active gastroesophageal flux disease (Amendment number 1)
* Concomitant treatment with analgesics or any other drug that may have influenced the headache symptomatology - including metamizol or ASA -, was referred to its use during the headache episodes under evaluation. As long as appropriate wash-out periods were respected, analgesics were allowed in between the episodes of tension headache (TH) and their use as a rescue medication did not lead to the exclusion of the patient (Amendment number 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 1998-10; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Time-interval weighted sum of pain intensity difference (SPID) on a Visual Analogue Scale (VAS) | before and 30 minutes, 1, 2, 3, and 4 hours after drug intake

SECONDARY OUTCOMES:
Pain intensity difference (PID) on a VAS | before and 30 minutes, 1, 2, 3, and 4 hours after drug intake
Maximum pain intensity difference (MAXPID) on a VAS | before and 30 minutes, 1, 2, 3, and 4 hours after drug intake
Number of patients with at least a 50% pain reduction on a VAS | before and 30 minutes, 1, 2, 3, and 4 hours after drug intake
Time to 50% pain intensity reduction on a VAS | before and 30 minutes, 1, 2, 3, and 4 hours after drug intake
Maximum pain relief (MAXPAR) on a Verbal Rating Scale (VRS) | 30 minutes, 1, 2, 3, and 4 hours after drug intake
Total pain relief (TOTPAR) on a VRS | 30 minutes, 1, 2, 3, and 4 hours after drug intake
Number of patients using rescue medication | 2, 3, and 4 hours after drug intake
Global efficacy assessment on a VRS by the patient and investigator | 4 hours after drug intake
Number of patients with adverse events | up to 2 months